CLINICAL TRIAL: NCT03637673
Title: The Possible Role of Thyroxine in Keratoconus Development
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Amir abou Samra, Dr., Alexandria University
Other Study IDs: 5621
Record Dates: First submitted 2018-08-15; First posted 2018-08-20 (Actual); Last update posted 2018-08-20 (Actual); Status verified 2018-08

CONDITIONS: Keratoconus
MeSH Terms: conditions — Keratoconus

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples to measure T3,T4, TSH level
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Keratoconus (KC) is a corneal ectatic disorders, with incidence rate 1 per 50,000 among the population. Hormonal imbalances may be associated with KC as it affects the corneal metabolism. In this study, we aim to examine this clinical association between thyroid gland dysfunction (TGD) and KC.

DETAILED DESCRIPTION:
Keratoconus (KC) is a corneal ectatic disorders, with incidence rate 1 per 50,000 among the population. Moreover, the pathophysiological processes underlying KC have not been fully elucidated with proposed mechanisms to include proteolytic degradation in the corneal stroma, oxidative damage, epithelial mechanical injury, immunological factors, and genetic factors. However, Hormonal imbalances may be associated with KC as it affects the corneal metabolism. Furthermore, thyroid gland dysfunction (TGD) can frequently associated with eye diseases such as Graves disease. Previous studies investigated the association between TGD and KC. Interestingly, thyroxine (T4) is important for corneal dehydration and transparency during embryonic development and regulates the synthesis of keratin sulfate proteoglycan in the chicken. T4 receptors (T4Rs) have been found in the lacrimal gland, confirming that the tear producing gland is a target organ of T4. T4 level was elevated in the tears of patients with KC. Hence, in this study, we aim to investigate the clinical association between TGD and KC.

ELIGIBILITY:
Inclusion Criteria:

* Patients with KC.

Exclusion Criteria:

* Patients who cannot give an informed consent.
* Patients who cannot provide needed samples for any reason

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We will enroll all patients who meet the inclusion criteria and signed a written informed consent form.
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2018-06-01 (Actual); Primary Completion 2018-08-30 (Estimated); Study Completion 2018-09-15 (Estimated)

PRIMARY OUTCOMES:
measuring the serum concentrations of free T4 (fT4) and thyroid-stimulating hormone (TSH) | We will recruit patients who meet the inclusion criteria during the study period of 3 months (June- August 2018). We will take only one blood sample from each patient recruited after the recrutiement and during this period
  The endocrinologic examination will include measuring the serum concentrations of free T4 (fT4) and thyroid-stimulating hormone (TSH) using an immunoassay method (ADVIA Centaur; Bayer Diagnostics, Germany). The normal reference ranges for TSH and fT4 were determined to be 0.35 to 4.5 mIU/ L and 0.7 to 1.65 ng/dL, respectively. Clinical cases with fT4 serum concentrations beyond these reference ranges will be defined as TGD. All examinations will be handled anonymously.

CONTACTS AND LOCATIONS:
Locations (1):
- Alexandria Faculty of Medicine, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No